CLINICAL TRIAL: NCT04984590
Title: Early Feasibility Study to Evaluate the Safety and Effectiveness of the Intraoperative Pseudophakic Capsular Lens Magnifier for Age-Related Macular Degeneration (IOPCL AMD-MAG) for Secondary Implantation in the Capsular Bag to Improve Near Vision in Subjects With Age-Related Macular Degeneration After Cataract Surgery
Brief Title: Early Feasibility Study Using IOPCL MAG to Improve Near Vision in ARMD Subjects
Status: Completed | Type: Interventional
Sponsor: OnPoint Vision Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOPCL AMD-20
Record Dates: First submitted 2021-07-13; First posted 2021-07-30 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Low Vision; Age Related Macular Degeneration
MeSH Terms: conditions — Vision, Low; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Treatment with IOPCL AMD MAG at least 6-months after cataract surgery with Alcon Model SN60WF or SA60AT
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- IOPCL AMD MAG (Other): All subjects will receive a 10.0 Diopter intraocular pseudophakic capsular lens magnifier (IOPCL MAG)
  Interventions: Device: IOPCL AMD MAG

INTERVENTIONS:
Device: IOPCL AMD MAG — The IOPCL MAG (intraocular pseudophakic capsular lens magnifier) consists of a 4.5 mm diameter optic. The central 1.8mm of the anterior surface has a power of 10.0 diopters. This IOPCL MAG will be implanted over an Alcon Model SN60WF or SA60AT intraocular lens to improve near vision.

SUMMARY:
This early feasibility study aims to improve near vision in subjects 55 years or older who have a clinical diagnosis of Age-Related Macular Degeneration. Subjects must have previously been implanted with either the Alcon Model SN60WF or Model SA60AT intraocular lens at least 6-months prior to receiving the IOPCL (intraocular pseudophakic capsular lens). Subject will be followed for a period of 12-months.

DETAILED DESCRIPTION:
This will be a 12-month study, in which a maximum of 10 pseudophakic subjects from up to three clinical sites with a diagnosis of age-related macular degeneration will be enrolled. The IOPCL MAG (intraocular pseudophakic capsular lens magnifier) consists of a 4.5mm diameter optic. The IOPCL MAG is centered above the existing intraocular lens. The IOPCL MAG is designed to improve near vision of the AMD subject by providing magnification of 10 diopters in the central 1.8mm zone of the lens optic.

The primary objective of this study is to determine the stability of the IOPCL-AMD-MAG to successfully adhere to a pseudophakic intraocular lens (PCIOL) without slippage or rotation.

The secondary objective of this study is to determine if the IOPCL-AMD-MAG can improve uncorrected near vision in subjects previously implanted with the Alcon Models SN60WF or SA60AT.

Outcome simulation testing will be performed prior to the subject receiving the IOPCL. To qualify for the study the subject must demonstrate an improvement in uncorrected near visual acuity of 10 letters over baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 55 years or older.
2. Subjects who have already had cataract surgery with an Alcon SN60WF or SA60AT monofocal intraocular lens with a lens power between 17.0 diopters and 24.0 diopters clearly evidenced by photographic documentation by one of the following:

   * patient medical record
   * clinic chart with labeling attached
   * surgical record with labeling attached, or
   * patient identification card with make, model and serial number.
3. Subjects who have already had cataract surgery at least 6 months from the planned date of the IOPCL surgery.
4. Subjects who have had a Nd: YAG capsulotomy at least 1 month prior to the planned date of the IOPCL surgery.
5. Subjects with non-neovascular dry AMD meeting the following criteria:

   * No change in Amsler Grid test within the past 12 months
   * No subretinal fluid or macular hemorrhage confirmed by optical coherence tomography (OCT) imaging.
   * No fundoscopic changes within the past 12 months (i.e., changes in retinal pigment epithelium).
6. Subjects with best corrected distance visual acuity from 20/80 to 20/800.
7. Subjects with a preoperative manifest refraction spherical equivalent (MRSE) of +1.0D to -1.0D.
8. Subjects with ≤1.0D of corneal cylinder determined by keratometry readings.
9. Subjects who are unsatisfied with their current near vision correction provided by either spectacles or external magnifier.
10. Subjects who demonstrate at least 10 letters of near visual acuity improvement with the simulation/tolerance test (using manifest refraction with +7.0D add) compared to conventional near vision testing (using manifest refraction with +3.0D add).
11. Subjects with a minimum endothelial cell count of 1800 cells/mm2.
12. Subjects willing to abstain from pursuing any other surgical vision-correcting procedures for the duration of the study.
13. Subjects who are willing and able to complete all required postoperative visits.
14. Subjects who are able to comprehend and sign a statement of informed consent.

Exclusion Criteria:

1. Subjects who have already had cataract surgery with a toric or multifocal or accommodating Intraocular Lens.
2. Subjects who have already had cataract surgery with an Alcon SN60WF or SA60AT monofocal intraocular lens with a power below 17.0 diopters and greater than 24.0 diopters.
3. Subjects with neovascular (wet) AMD.
4. Subjects who have not had an Nd: YAG capsulotomy.
5. Subjects who were treated with an IOL off-label.
6. Subjects who have more than 1.0D of corneal cylinder determined by Keratometry readings.
7. Subjects whose continuous curvilinear capsulorhexis was less than 5mm or more than 6.0 mm in size at the time of IOL surgery.
8. Subjects who had cataract surgery less than 6 months from the planned date of the IOPCL surgery.
9. Subjects with anterior capsule fibrosis and phimosis that in the opinion of the investigator may confound the outcome or increase the risk to the subject.
10. Subjects who do not gain at least 10 letters of near visual acuity with the simulation/tolerance testing (using manifest refraction with +7.0D add) compared to conventional near vision testing (using manifest refraction with +3.0D add).
11. Subjects with a concomitant retinal or choroidal disorder other than AMD.
12. Subjects with any corneal abnormality, other than regular corneal astigmatism that in the opinion of the investigator would confound the outcome(s) of the study.
13. Subjects with clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy).
14. Subjects with microphthalmos.
15. Subjects with a previous retinal detachment.
16. Subjects with a recurrent severe anterior or posterior segment inflammation of unknown etiology.
17. Subjects with iris neovascularization.
18. Subjects with glaucoma.
19. Subjects with advanced visual field defects (e.g., central large scotoma where magnification would not help).
20. Subjects with a fundus not visible.
21. Subjects with aniridia.
22. Subjects with advanced optic nerve atrophy.
23. Subjects with damaged or incomplete zonules.
24. Subjects with a known history of pseudoexfoliation.
25. Subjects with acute, chronic or uncontrolled systemic or ocular disease that in the opinion of the investigator would increase the operative risk or confound the outcome(s) of the study.
26. Subjects with medications that, in the opinion of the investigator, may confound the outcome or increase the risk to the subject (tamsulosin hydrochloride (Flomax)) or other medications with similar side effects (floppy iris syndrome).
27. Subjects with cognitive impairment that may interfere with the ability to understand the potentially complex considerations underlying an informed decision on trial participation and/or interfere with the ability to neuro-adapt to this device in the postoperative period.

    -

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | IOPCL AMD MAG
Started | 9; 9 Eyes
Completed | 9; 9 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.2 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not of Hispanic, Latino/a, or Spanish origin | 9
  White | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Tilt of the PCIOL and IOPCL MAG Complex
Description: Measuring postoperative tilt of the PCIOL and IOPCL MAG complex. Tilt was defined as less than or equal to 10 degrees.
Time Frame: 12 Months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  PCIOL Tilt <= 10 degrees | 9
  IOPCL MAG Tilt <=10 degrees | 9

2. Primary Outcome: IOPCL MAG Decentration
Description: Measures the decentration of the IOPCL MAG against the PCIOL. Decentration was defined as the horizontal and vertical distances greater than or equal to 0.25mm or less than or equal to 0.75mm.
Time Frame: 12 Months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Number of eyes with IOPCL MAG horizontal and vertical distances >= 0.25mm and <=0.75mm | 9
  Number of eyes with IOPCL MAG horizontal and vertical distances < 0.25mm and >0.75mm | 0

3. Primary Outcome: Uncorrected Near Visual Acuity at 14cm Change From Baseline (Letters) (≥ 75% Achieving ≥ 10 Letters)
Description: Proportion of eyes (≥ 75%) able to achieve improvement of 10 letters or more of uncorrected near visual acuity (at 14 cm) at 12 months from baseline
Time Frame: 12 Months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 8
  Gain of >= 15 letters (>= 3 lines) | 9
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >=10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>=3 lines) | 0

4. Secondary Outcome: Uncorrected Near Visual Acuity at 14cm Change From Baseline (Letters) (≥ 50% Achieving ≥ 20 Letters)
Description: Proportion of eyes (≥ 50%) able to achieve improvement of 20 letters or more of uncorrected near visual acuity (at 14 cm) at 12 months from baseline
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 8
  Gain of >= 15 letters (>= 3 lines) | 9
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >= 10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>= 3 lines) | 0

5. Secondary Outcome: Postoperative Uncorrected Near Visual Acuity at 14cm Compared to Preoperative Best Corrected Near Visual Acuity at 30cm With +3.0D Add (≥ 75% Achieving ≥ 10 Letters)
Description: Proportion of eyes (≥ 75%) able to achieve improvement of 10 letters or more when comparing uncorrected near visual acuity (UCNVA) (at 14 cm) at 12 months from baseline BCNVA (at 30 cm, wearing the appropriate preoperative distance refractive correction in addition to +3.0D add)
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 5
  Gain of >= 15 letters (>= 3 lines) | 8
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >= 10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>= 3 lines) | 0

6. Secondary Outcome: Postoperative Uncorrected Near Visual Acuity at 14cm Compared to Preoperative Best Corrected Near Visual Acuity at 30cm With +3.0D Add (≥ 50% Achieving ≥ 20 Letters)
Description: Proportion of eyes (≥ 50%) able to achieve improvement of 20 letters or more when comparing uncorrected near visual acuity (UCNVA) (at 14 cm) at 12 months from baseline BCNVA (at 30 cm, wearing the appropriate preoperative distance refractive correction in addition to +3.0D add)
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 5
  Gain of >= 15 letters (>= 3 lines) | 8
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >= 10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>= 3 lines) | 0

7. Secondary Outcome: Postoperative Best Corrected Near Visual Acuity at 14cm Compared to Preoperative Best Corrected Near Visual Acuity at 30cm With +3.0D Add (≥ 75% Achieving ≥ 10 Letters)
Description: Proportion of eyes (≥ 75%) able to achieve improvement of 10 letters or more when comparing best corrected near visual acuity (BCNVA) (at 14 cm) at 12 months from baseline BCNVA (at 30 cm, wearing the appropriate preoperative distance refractive correction in addition to +3.0D add)
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 5
  Gain of >= 15 letters (>= 3 lines) | 8
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >= 10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>= 3 lines) | 0

8. Secondary Outcome: Postoperative Best Corrected Near Visual Acuity at 14cm Compared to Preoperative Best Corrected Near Visual Acuity at 30cm With +3.0D Add (≥ 50% Achieving ≥ 20 Letters)
Description: Proportion of eyes (≥ 50%) able to achieve improvement of 20 letters or more when comparing best corrected near visual acuity (BCNVA) (at 14 cm) at 12 months from baseline BCNVA (at 30 cm, wearing the appropriate preoperative distance refractive correction in addition to +3.0D add)
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IOPCL AMD MAG
Number analyzed (Participants) | 9
Number analyzed (Eyes) | 9
Eyes
  Gain of >= 20 letters (>= 4 lines) | 5
  Gain of >= 15 letters (>= 3 lines) | 8
  Gain of >= 10 letters (>= 2 lines) | 9
  Gain of >= 5 letters (>= 1 line) | 9
  No change | 0
  Loss of >= 5 letters (>= 1 line) | 0
  Loss of >= 10 letters (>= 2 lines) | 0
  Loss of >= 15 letters (>= 3 lines) | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | IOPCL AMD MAG
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOPCL AMD MAG (N=9)
Bilateral pruritis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04984590/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04984590/SAP_001.pdf